CLINICAL TRIAL: NCT01937884
Title: Supplemental Parenteral Nutrition in Pediatric Respiratory Failure
Acronym: SuPPeR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll patients
Sponsor: University of Arizona (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Katri Typpo, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-0374; 5K12HD047349-09 (NIH)
Record Dates: First submitted 2013-09-01; First posted 2013-09-10 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Acute Respiratory Failure With Hypoxia; Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Parenteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Parenteral Nutrition (Experimental): Patients receive supplemental parenteral nutrition within 12 hours of enrollment. Titrated with enteral nutrition to achieve target goal calories and protein.
  Interventions: Drug: Parenteral Nutrition
- Late Parenteral Nutrition (Active Comparator): Patients receive supplemental parenteral nutrition 96 hours after enrollment. Titrated with enteral nutrition to achieve target goal calories and protein.
  Interventions: Drug: Parenteral Nutrition

INTERVENTIONS:
Drug: Parenteral Nutrition

SUMMARY:
Optimal delivery of nutritional support during critical illness is central to appropriate intensive care unit management, and yet fundamental gaps in knowledge exist regarding timing, route, dose, and type of nutritional support for critically ill infants and children. Understanding how to optimize nutritional support during pediatric critical illness is important because even brief periods of malnutrition in infancy result in permanent negative effects on long-term neurocognitive development. Optimized nutrition support is a way to improve morbidity for survivors of pediatric critical illness. Parenteral nutrition (PN) supplementation could improve long-term neurocognitive outcome for pediatric critical illness by preventing acute malnutrition, but has unknown effects on intestinal barrier function; a proposed mechanism for late sepsis and infectious complications during critical illness.

While randomized controlled trials (RCT) support early PN in premature infants and late PN in critically ill adults, the optimal time to begin PN is unknown for critically ill infants and children. Acute malnutrition may develop within 48 hours of admission in critically ill infants and children, and repleted energy stores are predictive of survival. And yet, due to concerns for PN-associated infectious morbidity, current PICU standard of care is to supplement with PN only in children who fail to enterally feed, as late as 7 days into their admission. Delays in nutrition may have long-term effects on cognitive outcome in older infants and children. In premature infants, PN begun within hours of birth results in improved 18-month neurocognitive outcome without an increase in infectious complications. An RCT is needed to determine if early PN in critically ill infants and children prevents acute malnutrition and improves short and long-term outcomes of PICU hospitalization.

The central hypothesis of this proposal is that optimized early protein and calorie delivery will improve nutritional outcomes and intestinal barrier function for critically ill infants and children. The overall purpose of this study is to evaluate the efficacy and safety of early PN as a supplement to enteral nutrition to improve nutritional delivery, nutritional outcomes, and intestinal barrier function for infants and children with acute respiratory failure who are mechanically ventilated in the pediatric intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to study hospital pediatric intensive care unit (PICU),
2. One month to 16 years of age,
3. Exhibits Acute Hypoxemic Respiratory Failure as defined as: PaO2/FiO2 ≤ 300 or SpO2/FiO2 ≤ 260, No evidence of cardiac dysfunction, Mechanically ventilated,
4. Require artificial nutrition,
5. Anticipate placement of central venous line within 24 hours of admission

Exclusion Criteria:

1. Premature infants and neonates < 37 weeks corrected gestational age,
2. Transfer patient on an established enteral or parenteral nutritional regimen,
3. Known allergy to lactulose or mannitol,
4. Pregnant,
5. Admit BMI >30,
6. Thoracic trauma, abdominal trauma, and/or active intracranial bleeding,
7. Anuric renal failure, previous bowel surgery and/or short gut syndrome,
8. Cannot be enterally fed within 24 hours of admission according to the admitting physician,
9. On extracorporeal membrane oxygenation (ECMO),
10. Expected survival <24 hours or limitations to aggressive ICU care (DNR),
11. Receiving active CPR when admitted to the PICU,
12. A pre-existing bronchopleural fistula,
13. Previously enrolled and randomized into this protocol,
14. Actively enrolled in another clinical trial which at the discretion of the PI would conflict with this study.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katri V Typpo, MD, MPH, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Parenteral Nutrition: Patients receive supplemental parenteral nutrition within 12 hours of enrollment. Titrated with enteral nutrition to achieve target goal calories and protein over the one week study period.
- Late Parenteral Nutrition: Patients receive supplemental parenteral nutrition 96 hours after enrollment if meeting < 80% of caloric goals with enteral nutrition alone. Titrated with enteral nutrition to achieve target goal calories and protein over the one week study period.
Period: Overall Study
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Started | 7 | 11
Completed | 6 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 1.4 [0.4 to 4.3] | 1.1 [0.4 to 6.0] | 1.3 [0.4 to 4.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
BMI z score [Median (Inter-Quartile Range); unit: Z score] — The BMI Z-Score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. BMI Z-score cut-points of < - 2.0, > 1.0, > 2.0, > 3.0 define wasted, at risk of overweight, overweight and obese, respectively. BMI z scores were calculated used CDC growth charts for children 2 years of age and older. For children under 2 years of age the weight for age Z score is reported.
  Z score | -.73 [-1.7 to 0.2] | -.9 [-1.2 to -0.03] | -0.9 [-1.7 to 0.21]
PELOD-2 score [Median (Inter-Quartile Range); unit: units on a scale] — The Pediatric Logistic Organ Dysfunction-2 (PELOD-2) score allows assessment of the severity of organ dysfunction on a continuous scale. The score incorporates assessment of 5 organ system dysfunction (Cardiovascular, Neurologic, Respiratory, Hematologic, and Renal). Component scores for each organ system can be calculated, only the composite score which reflects baseline severity of illness and organ dysfunction is reported in our study. The minimum PELOD-2 score is 0 and the maximum is 33. A higher PELOD-2 score indicates a higher probability of death.
  units on a scale | 8 [6 to 9] | 7 [5 to 9] | 7.5 [6 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Modified Prognostic Inflammatory and Nutritional Index (PINI)
Description: The change day 0 to day 5 of the modified Prognostic Inflammatory and Nutritional Index (PINI) is a quantitative method to monitor the relation between markers of nutrition and acute phase proteins. It allows assessment of nutrition markers in the context of acute inflammation and in response to early enteral nutrition. A higher baseline PINI score indicates higher degree of inflammation. The modified PINI is calculated by the the ratio of (C-Reactive Protein(mg/dL) x Fibrinogen (mg/dL))/ (Transferrin (mg/dL) x Transthyretin (mg/dL)). The average change in the modified PINI from day 0 to day 5 critically ill children receiving early enteral nutrition is a decrease by 5.3 +/- 3.2 (mean +/- standard error of the mean) (Briassoulis et.al. Nutrition 2001). A larger negative number for the change from day 0 to day 5 indicates a greater degree of inflammation resolution.
Time Frame: Change in PINI from day 0 to day 5
Population: Patients with central venous access and/or arterial access removed at study day 5 did not have blood drawn for PINI measurement. All patients with paired PINI values from day 0 and day 5 obtained are analyzed based on initial group assignment.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Early Parenteral Nutrition: Patients receive supplemental parenteral nutrition within 12 hours of enrollment. Titrated with enteral nutrition to achieve target goal calories and protein.
  Parenteral Nutrition
- Late Parenteral Nutrition: Patients receive supplemental parenteral nutrition 96 hours after enrollment. Titrated with enteral nutrition to achieve target goal calories and protein.
  Parenteral Nutrition
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Number analyzed (Participants) | 4 | 7
score on a scale | -1.6 (1.0) | -3.2 (1.8)
Statistical Analysis 1: Comparison: Early Parenteral Nutrition vs Late Parenteral Nutrition; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Cumulative Percent of Daily Goal Calories Achieved
Description: Evaluate percentage of cumulative goal calories achieved through parenteral and enteral routes in both study arms until patient exits study participation. Measure is calculated by (sum of kcal delivered over days of study participation/number of days in study).
Time Frame: baseline and daily through day 7
Population: All patients enrolled had daily nutrition data collected until end of study participation.
Measure: Median (Inter-Quartile Range); unit: percent of goal kcal/day
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Number analyzed (Participants) | 7 | 11
percent of goal kcal/day | 103.8 [98.5 to 110.2] | 103.4 [86.4 to 110.0]
Statistical Analysis 1: Comparison: Early Parenteral Nutrition vs Late Parenteral Nutrition; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Plasma Intestinal Fatty Acid Binding Protein (I-FABP)
Description: The percent change in plasma Intestinal Fatty Acid Binding Protein from baseline to study day 5, prior to late PN initiation
Time Frame: baseline and day 5
Population: All patients enrolled in the study with IFABP results obtained at baseline and hour 96, analyzed in initial assigned groups.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Number analyzed (Participants) | 5 | 8
percent change | 2.11 [-35.9 to 28.3] | -25 [-47.9 to 8.6]
Statistical Analysis 1: Comparison: Early Parenteral Nutrition vs Late Parenteral Nutrition; Test type: Superiority; p = 0.27, t-test, 2 sided; Student's t-test on log-transformed change in IFABP

4. Secondary Outcome: Plasma Citrulline
Description: Evaluates absolute plasma citrulline concentration as a measure of functional enterocyte mass. A higher citrulline concentration indicates a higher functional enterocyte mass. Healthy children have an average citrulline concentration of 25 +/- 9 uMol/L. Assessed on day 0 and day 5, results reported for day 0 and 5. Outcome analysis on difference between treatment groups on day 5.
Time Frame: baseline and day 5
Population: Citrulline concentrations obtained for patients with plasma samples available for analysis on study day 0 and 5
Measure: Median (Inter-Quartile Range); unit: umoL per Liter
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Number analyzed (Participants) | 7 | 11
umoL per Liter
  day 0 | 10 [8.6 to 14.8] | 8 [4.7 to 11]
  day 5: number analyzed (Participants) | 5 | 8
  day 5 | 19.4 [19 to 32.5] | 14.5 [11.1 to 20.4]
Statistical Analysis 1: Comparison: Early Parenteral Nutrition vs Late Parenteral Nutrition; Test type: Superiority; p = 0.04, t-test, 2 sided; Student's t-test on log-transformed citrulline concentration on study day 5, by treatment group

5. Secondary Outcome: Plasma Claudin 3
Description: As a measure of enterocyte tight junctions, calculate the percent change in plasma claudin 3 concentrations from baseline (day 0) and study day 5, prior to late PN administration.
Time Frame: baseline through hour 96
Population: Included all patients with claudin 3 plasma concentrations reported at hour zero and 96, analyzed in groups as initially assigned.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Number analyzed (Participants) | 5 | 8
percent change | 29.8 [11.7 to 53.6] | 111.7 [-8.8 to 224.1]
Statistical Analysis 1: Comparison: Early Parenteral Nutrition vs Late Parenteral Nutrition; Test type: Superiority; p = 0.43, t-test, 2 sided; Student's t-test on log-transformed percent change of claudin 3

6. Secondary Outcome: Gastrointestinal Permeability
Description: Gastrointestinal permeability measured with the ratio of urinary recovery of lactulose and mannitol on day 5 of study participation. The range of values is generally reported as 0.02 to 2.2 with a higher value indicating greater gastrointestinal permeability. Values obtained on day 0 and day 5, day 5 reported.
Time Frame: day 5
Population: Analysis of lactulose and mannitol urinary concentrations performed on all patients who received the lactulose and mannitol study test and with urinary samples obtained on day 5.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Number analyzed (Participants) | 5 | 8
ratio | 0.15 [0.13 to 0.78] | 0.17 [0.13 to 0.24]
Statistical Analysis 1: Comparison: Early Parenteral Nutrition vs Late Parenteral Nutrition; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Number of Participants With Hospital-Acquired Infections
Description: Record any hospital-defined hospital acquired infections through day 28 in all study participants.
Time Frame: until hospital discharge or day 28 if still hospitalized
Population: All study participants
Measure: Count of Participants; unit: Participants
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Number analyzed (Participants) | 7 | 11
Participants | 0 | 1
Statistical Analysis 1: Comparison: Early Parenteral Nutrition vs Late Parenteral Nutrition; Test type: Superiority; p = 0.43, Chi-squared

8. Other Pre Specified Outcome: 28-day Mortality
Description: Death of a study patient do to any cause measured up to 28 days after study enrollment.
Time Frame: 28 days
Population: Determined for all study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
Number analyzed (Participants) | 7 | 11
Participants | 2 | 0
Statistical Analysis 1: Comparison: Early Parenteral Nutrition vs Late Parenteral Nutrition; Test type: Superiority; p = 0.06, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 14 days, from time of patient enrollment
Description: Adverse event reporting follows the clinicaltrials.gov definitions and includes all-cause mortality, serious adverse events, and other adverse events.
Arm/Group | Early Parenteral Nutrition | Late Parenteral Nutrition
All-Cause Mortality (participants affected / at risk) | 2/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 5/11
Other Adverse Events (participants affected / at risk) | 5/7 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Parenteral Nutrition (N=7) | Late Parenteral Nutrition (N=11)
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 3 (3) — Identification of a deep vein thrombosis by ultrasound imaging
Hospital-Acquired infection (Infections and infestations) | 0 (0) | 1 (1) — Hospital-determined hospital acquired infections
Aspiration of gastric contents (Gastrointestinal disorders) | 0 (0) | 1 (1) — Aspiration event as determined by the Clinical team
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Parenteral Nutrition (N=7) | Late Parenteral Nutrition (N=11)
Desaturation < 85% (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 5 (9) — Desaturation event with SaO2 < 85%
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Glucose value >200 mg/dL

LIMITATIONS AND CAVEATS:
This study was discontinued early due to slow enrollment. The small study size limits interpretation of clinical and biochemical outcomes data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT01937884/Prot_SAP_000.pdf